CLINICAL TRIAL: NCT02681588
Title: Impact of Maternal Obesity on Fetal Development and Perinatal Events. Analysis of the Determinants of Fetal Growth.
Brief Title: Newborns of Obese Mothers
Acronym: MOBENN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P081109
Record Dates: First submitted 2016-02-10; First posted 2016-02-12 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-02

CONDITIONS: Obesity
Keywords: diabetes, obesity, skinfold, newborn
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Obese group (Experimental)
  Interventions: Procedure: Obstetric management
- Normal Weight group (Active Comparator)
  Interventions: Procedure: Obstetric management

INTERVENTIONS:
Procedure: Obstetric management — Screening for gestational diabetes at 32 weeks of gestation, determination of fasting glucose during late pregnancy ; blood samples on arrival at the delivery room ; drawing blood from the umbilical cord after section; skinfold measurement of the newborn within 72 hours of life.

SUMMARY:
This was a prospective bi-centric study, exposed-unexposed. In an effort to better understand the potential independent effect of maternal obesity on fetal growth, investigators designed a prospective study, comparing fetal growth between normal weight (18.5 ≤ BMI < 25 kg/m2) or obese pregnant women (BMI ≥ 30 kg/m2), while maternal diabetes and hyperglycaemia was screened and treated throughout pregnancy.

DETAILED DESCRIPTION:
The study population concerned obese pregnant women (BMI ≥ 30 kg / m² before pregnancy) and their newborn and normal weight pregnant women (18.5 ≤IMC <25 kg/m²) and their newborn as control. Inclusion criteria were body mass index (BMI) ≥ 30 kg/m2 or 18.5 ≤ BMI < 25 kg/m2, 18 ≤ age ≤ 40 years, singleton pregnancy. Exclusion criteria were: 25 ≤ BMI <30 kg/m2, age < 18 or > 40 years, multiple pregnancy, first consultation after 18 WG, pregestational diabetes, obesity due to genetic disorder or secondary to intracranial tumor or radiotherapy, bariatric surgery, chronic diseases other than the obesity, inability to converse in French language. The matching criteria for controls were: age ± 5 years, primigravida or multigravida, duration of gestation ± 4 weeks.

The main objective of this project was to assess the independent effect of maternal obesity:

* on the weight and adipose tissue of newborn
* on the function of adipose tissue (production of leptin and adiponectin)
* on fetal growth factors (C-peptide, IGF-1)
* on carbohydrate metabolism of the newborn. Two maternities were involved in the study: Pitié Salpêtrière and Armand Trousseau, in Paris, France. This research was conducted over a 3 years period. The duration of participation of each woman corresponded to the duration of pregnancy care and duration of care for the newborn immediately after birth, usually the length of stay in the maternity.

The only differences compared to the usual care included:

* Additional oral glucose tolerance test at 32 weeks of gestation;
* Determination of fasting blood glucose during late pregnancy
* Maternal blood samples on arrival at the delivery room
* Drawing blood from the umbilical cord after section;
* Skinfold measurement of the newborn within 72 hours of life.

ELIGIBILITY:
Inclusion Criteria:

1. - BMI ≥30 kg / m² or between 18.50 and 24.99 kg / m².
2. - Pregnant woman coming to the centre before 18 weeks of gestation.
3. - Age ≥ 18 and ≤ 40 years
4. - Single Pregnancy
5. - No constitutional or progressive disease other than obesity: inflammatory disease, epilepsy, pathology psychiatric, tumor...
6. - Informed written consent.

Exclusion Criteria:

1. - Pregnant woman coming to the center after 18 weeks of gestation, BMI <18.5 kg / m² or between 25 and 29.99 Kg / m².
2. - Age <18 or> 40 years
3. - Multiple pregnancy
4. - Presence of a constitutional disease or progressive disease other than obesity.
5. - Patients who underwent obesity surgery type "bypass" or gastroplasty
6. - Obesity secondary to genetic disorder, intracranial lesions or pituitary radiotherapy
7. - not stabilized endocrine pathology.
8. - pregestational diabetes
9. - No affiliation to a social security scheme

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 496 (Actual)
Dates: Start 2010-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
ponderal index measured by a balance | at birth
skinfold's measure measured by a special clamp | at birth
birthweight | at birth